CLINICAL TRIAL: NCT04426318
Title: COVID-19 and the Healthy Minds Program for Educators
Acronym: CAHMP-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Chan Zuckerberg Initiative (Other); Healthy Minds Innovations (Other); Center for Healthy Minds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0533; A171600 (Other: UW Madison); EDUC/COUNSELING PSYCH (Other: UW Madison); Protocol Approval 10/15/2020 (Other: UW Madison)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Depression; Psychological Stress; Psychological Distress; Well-being
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological | interventions — Meditation; Mindfulness

STUDY DESIGN:
Intervention Model Description: Random parallel assignment
Who Masked: Investigator
Masking Description: There is no outcome assessor - all assessments will be conducted online by participants. Investigators will be blind to group assignment during data analysis. Analysis of hypotheses related to baseline characteristics, adherence and dosage cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Minds Program Foundations Training (Experimental): Healthy Minds Program (HMP) Description:
  The HMP app was developed by Healthy Minds Innovations at the UW Center for Healthy Minds, and is based on the work of Richard Davidson, PhD. HMP is designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of high-quality guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). HMP has >100 guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
  Interventions: Behavioral: Healthy Minds Program Foundations Training
- Wait-list control (No Intervention): Participants assigned to the wait-list control will not receive treatment for the intervention and follow-up period. They will be provided access to the HMP Foundations training after completing follow-up testing.

INTERVENTIONS:
Behavioral: Healthy Minds Program Foundations Training — The HMP is a novel, smartphone-based app that provides a series of guided meditation practices on four primary constituents of well-being: Awareness, Connection, Insight, and Purpose. The program is unique in several ways. First, all program elements are introduced with a summary of the scientific evidence supporting its constituent elements (e.g., Awareness and well-being). Second, in addition to standard sitting meditation practices found in many meditation-based behavioral interventions, the HMP offers active practices in which participants can develop the same skills but while embedding practice into activities they already do in their normal daily routine.
  Other Names: meditation; mindfulness
  Arms: Healthy Minds Program Foundations Training

SUMMARY:
This study is a randomized controlled trial (RCT) of the four-week Healthy Minds Program (HMP) app Foundations training in employees of a mid-size urban school district in the United States during the summer of 2020, in the midst of the novel coronavirus pandemic. A 3-month follow-up in the fall of 2020 will also be conducted.

Participants will be recruited via email and mailed postcards, and will first complete an online screen. Eligible participants will then enter a waiting zone for between 2-days and 2-weeks before they are sent the online pre-test. Upon completion of the pre-test, participants will be assigned to condition via a simple random number generator. If assigned to the intervention (i.e., the Healthy Minds Program App), participants will receive instructions and support in downloading and activating the app. Every 7-days over the 4-week intervention period participants in both conditions will complete the same set of measures. A full battery of measures will be administered a second time post-test, following the 4-week intervention period. Three-months after post-test, a follow-up assessment will be conducted.

The investigators predict that participants assigned to the intervention will demonstrate significantly reduced psychological distress after the intervention, and these decreases will persist at the 3-month follow-up. Further, it is hypothesized that baseline participant characteristics and early experience of the intervention will predict treatment adherence, study drop-out and outcomes, and that treatment engagement will moderate outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years old and up
* Employees of a K-12 school district in Wisconsin
* Smartphone or device that can download apps from Google Play or the iTunes app store

Exclusion Criteria:

* Individuals under 18 years old
* Significant meditation experience:

  1. Meditation retreat experience (meditation retreat or yoga/body practice retreat with significant meditation component),
  2. Regular meditation practice weekly for over 1 year OR daily practice within the previous 6 months; or
  3. Previous use of the HMP app.
* Patient-Reported Outcomes Measurement Information System (PROMIS) depression score > 70

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and listed in public data registries (i.e., osf) based on the publication of preregistered study hypotheses on a manuscript by manuscript basis.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be de-identified and made publicly available based on the publication of preregistered study hypotheses following peer review.
Access Criteria: Researcher consent. Any reasonable request will be granted.

REFERENCES:
- [Result] Goldberg SB, Baldwin SA, Riordan KM, Torous J, Dahl CJ, Davidson RJ, Hirshberg MJ. Alliance With an Unguided Smartphone App: Validation of the Digital Working Alliance Inventory. Assessment. 2022 Sep;29(6):1331-1345. doi: 10.1177/10731911211015310. Epub 2021 May 18. PMID 34000843
- [Result] Hirshberg MJ, Davidson RJ, Goldberg SB. Educators Are Not Alright: Mental Health During COVID-19. Educ Res. 2023 Jan;52(1):48-52. doi: 10.3102/0013189X221142595. PMID 37379444
- [Derived] Goldberg SB, Bolt DM, Dahl CJ, Davidson RJ, Hirshberg MJ. Does it matter how meditation feels? An experience sampling study. J Consult Clin Psychol. 2024 Aug;92(8):531-541. doi: 10.1037/ccp0000857. PMID 39347788
- [Derived] Webb CA, Hirshberg MJ, Gonzalez O, Davidson RJ, Goldberg SB. Revealing subgroup-specific mechanisms of change via moderated mediation: A meditation intervention example. J Consult Clin Psychol. 2024 Jan;92(1):44-53. doi: 10.1037/ccp0000842. Epub 2023 Sep 28. PMID 37768631
- [Derived] Webb CA, Hirshberg MJ, Davidson RJ, Goldberg SB. Personalized Prediction of Response to Smartphone-Delivered Meditation Training: Randomized Controlled Trial. J Med Internet Res. 2022 Nov 8;24(11):e41566. doi: 10.2196/41566. PMID 36346668
- See also: OSF Registry — https://osf.io/eqgt7

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8321 Wisconsin school system employees invited, 1136 self-screened for eligibility, 353 ineligible (for prior medication, prior HMP app use, or depression t-score greater than 70), 698 consented, 32 did not complete a pre-test, 666 assigned to an arm.
Groups:
- Healthy Minds Program Foundations Training: Healthy Minds Program (HMP) is a novel, smartphone-based app that provides a series of guided meditation practices on four primary constituents of well-being: Awareness, Connection, Insight, and Purpose. All program elements are introduced with a summary of the scientific evidence supporting its constituent elements (e.g., Awareness and well-being). In addition to standard sitting meditation practices found in many meditation-based behavioral interventions, the HMP offers active practices in which participants can develop the same skills but while embedding practice into activities they already do in their normal daily routine.
Period: Overall Study
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Started | 346 | 320
Failed Attention Checks | 4 | 6
Downloaded HMP App | 329 | 0
Completed T2 Assessment | 281 | 280
Completed T3 Assessment | 261 | 274
Completed T4 Assessment | 261 | 275
Completed T5 Assessment | 284 | 293
Completed T6 Assessment | 286 | 293
Final Intent to Treat Sample | 344 | 318
Completed | 344 | 318
Not Completed | 2 | 2
Not completed — failed attention checks and had their data removed from analyses | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control | Total
Number analyzed (Participants) | 344 | 318 | 662
Age, Customized [Count of Participants; unit: Participants]
  under 20 years | 0 | 1 | 1
  20-30 years | 55 | 46 | 101
  30-40 years | 105 | 90 | 195
  40-50 years | 103 | 93 | 196
  50-60 years | 61 | 79 | 140
  over 60 years | 20 | 9 | 29
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants were permitted to select more than one category.
  Participants
    Female | 302 | 281 | 583
    Male | 42 | 37 | 79
    Non-Binary | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaskan Native | 5 | 4 | 9
  Asian / Pacific Islander | 9 | 4 | 13
  Black / African American | 11 | 15 | 26
  Hispanic / Latino | 15 | 17 | 32
  White / Caucasian | 315 | 287 | 602
Region of Enrollment [Number; unit: participants]
  United States | 344 | 318 | 662
Highest Level of Education [Count of Participants; unit: Participants]
  less than 7 years formal education | 1 | 2 | 3
  Graduated High School | 10 | 6 | 16
  Some College | 24 | 27 | 51
  Graduated College | 100 | 103 | 203
  Advanced Degree | 208 | 178 | 386
  NA | 1 | 2 | 3
Household Income [Count of Participants; unit: Participants]
  Less than $20,000 | 8 | 9 | 17
  $20,000 - $40,000 | 22 | 19 | 41
  $40,000 - $70,000 | 80 | 82 | 162
  $70,000 - $100,000 | 87 | 74 | 161
  $100,000 - $200,000 | 135 | 121 | 256
  greater than $200,000 | 9 | 12 | 21
  Unknown | 3 | 1 | 4
Employment Category [Count of Participants; unit: Participants]
  Classroom Teacher | 144 | 134 | 278
  Classroom Support | 47 | 44 | 91
  Special Education Teacher | 29 | 31 | 60
  School Support | 38 | 35 | 73
  School Administrator | 8 | 4 | 12
  System Staff | 20 | 27 | 47
  Other / Unknown | 58 | 43 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on an Aggregate Measure of Psychological Distress That Averages the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety and Depressive Measures and the NIH Perceived Stress Scale
Description: Psychological distress will be assessed by aggregating 3 measures: PROMIS anxiety and PROMIS depression, and the NIH Toolbox Perceived Stress Scale. Averages will be z-scored with a mean of 0 and a standard deviation 1. Higher scores indicate increased psychological distress.
Time Frame: baseline, after weeks 1, 2, and 3 of the intervention, 4 weeks (post intervention), 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
z-score
  Baseline: number analyzed (Participants) | 342 | 315
  Baseline | 0.00 (0.88) | 0.00 (0.91)
  Week 1: number analyzed (Participants) | 277 | 276
  Week 1 | -0.29 (0.89) | -0.10 (0.95)
  Week 2: number analyzed (Participants) | 257 | 270
  Week 2 | -0.40 (0.85) | -0.10 (1.01)
  Week 3: number analyzed (Participants) | 257 | 271
  Week 3 | -0.55 (0.88) | -0.14 (1.02)
  Week 4: number analyzed (Participants) | 280 | 289
  Week 4 | -0.67 (0.89) | -0.20 (1.03)
  Week 16: number analyzed (Participants) | 282 | 289
  Week 16 | -0.55 (0.87) | -0.24 (1.00)

2. Secondary Outcome: Change From Baseline on the Five Facet Mindfulness Questionnaire Act With Awareness Subscale
Description: A measure of acting with mindful awareness. The total possible range in scores is 8-40, with higher scores indicating greater levels of this facet of mindfulness.
Time Frame: as for outcome 1
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 342 | 315
  baseline | 24.80 (5.93) | 24.56 (6.12)
  Week 1: number analyzed (Participants) | 277 | 276
  Week 1 | 24.19 (5.62) | 25.57 (6.15)
  Week 2: number analyzed (Participants) | 259 | 270
  Week 2 | 25.71 (5.47) | 25.69 (6.44)
  Week 3: number analyzed (Participants) | 258 | 271
  Week 3 | 26.45 (5.61) | 26.15 (6.21)
  Week 4: number analyzed (Participants) | 280 | 289
  Week 4 | 27.12 (5.67) | 26.12 (6.76)
  Week 16: number analyzed (Participants) | 282 | 290
  Week 16 | 27.1 (5.32) | 26.02 (6.36)

3. Secondary Outcome: Change From Baseline on the Drexel Defusion Scale (DDS)
Description: Psychological distancing (i.e., defusion) will be assessed with the 10-item Drexel Defusion Scale (DDS). The total possible range in scores is 0-50, with higher scores indicating greater levels of psychological distancing.
Time Frame: as for outcome 1
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 342 | 315
  baseline | 24.83 (7.89) | 24.45 (8.23)
  Week 1: number analyzed (Participants) | 276 | 275
  Week 1 | 27.14 (8.72) | 26.26 (8.31)
  Week 2: number analyzed (Participants) | 257 | 270
  Week 2 | 28.45 (8.42) | 26.96 (8.73)
  Week 3: number analyzed (Participants) | 255 | 270
  Week 3 | 29.61 (8.73) | 27.52 (9.07)
  Week 4: number analyzed (Participants) | 280 | 289
  Week 4 | 31.43 (8.54) | 27.92 (8.63)
  Week 16: number analyzed (Participants) | 281 | 289
  Week 16 | 30.93 (8.69) | 28.23 (8.57)

4. Secondary Outcome: Change From Baseline on the Meaning in Life Questionnaire
Description: The Meaning in Life Questionnaire Presence subscale will be used to measure perceptions of meaning and purpose in life. The total possible range in scores is 5 - 35 with higher scores indicating greater levels of meaning.
Time Frame: as for outcome 1
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 342 | 315
  baseline | 26.20 (5.44) | 25.81 (5.46)
  Week 1: number analyzed (Participants) | 278 | 276
  Week 1 | 26.83 (5.13) | 26.02 (5.38)
  Week 2: number analyzed (Participants) | 259 | 270
  Week 2 | 27.15 (5.14) | 25.85 (5.68)
  Week 3: number analyzed (Participants) | 258 | 271
  Week 3 | 27.62 (4.92) | 26.13 (5.83)
  Week 4: number analyzed (Participants) | 280 | 289
  Week 4 | 27.85 (5.35) | 26.02 (6.07)
  Week 16: number analyzed (Participants) | 282 | 290
  Week 16 | 27.91 (5.14) | 26.29 (5.87)

5. Secondary Outcome: Change From Baseline on the NIH Toolbox Loneliness Scale
Description: A measure of loneliness (i.e, lack of social connectedness). The total possible range in scores is 1-5, representing the average across all items; higher scores indicate greater levels of loneliness.
Time Frame: as for outcome 1
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 342 | 315
  baseline | 2.53 (0.77) | 2.58 (0.77)
  Week 1: number analyzed (Participants) | 278 | 276
  Week 1 | 2.34 (0.75) | 2.49 (0.74)
  Week 2: number analyzed (Participants) | 260 | 272
  Week 2 | 2.16 (0.72) | 2.38 (0.72)
  Week 3: number analyzed (Participants) | 259 | 271
  Week 3 | 2.02 (0.68) | 2.37 (0.75)
  Week 4: number analyzed (Participants) | 279 | 289
  Week 4 | 2.07 (0.71) | 2.33 (0.81)
  Week 16: number analyzed (Participants) | 283 | 291
  Week 16 | 2.13 (0.75) | 2.38 (0.82)

6. Secondary Outcome: Conway COVID Questionnaire Subscale Scores
Description: The Conway COVID Questionnaire is a new, 16-tem measure of coronavirus related distress and related experiences. Subscales include: perceived threat, financial scale, resource scale, psychological scale, symptoms scale, proximity to others scale, and news scale. Ratings from 1 to 7 with 1 = "not true of me at all" and 7 = "very true of me" with higher scores representing greater perceived threat. Mean for each subscale reported.
Time Frame: baseline
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 342 | 315
score on a scale
  Financial Subscale | 3.09 (2.08) | 3.00 (2.02)
  News Subscale | 4.03 (1.65) | 4.10 (1.55)
  Proximity Subscale | 3.16 (1.70) | 2.99 (1.66)
  Psychological Subscale | 4.45 (1.45) | 4.39 (1.44)
  Resource Subscale | 2.13 (1.85) | 2.00 (1.28)
  Symptoms Subscale | 1.65 (1.10) | 1.70 (1.17)
  Threat Subscale | 5.05 (1.35) | 5.03 (1.30)

7. Secondary Outcome: Conway COVID Questionnaire Subscale Scores
Description: as for outcome 6
Time Frame: 4 weeks (post intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 280 | 289
score on a scale
  Financial Subscale: number analyzed (Participants) | 279 | 289
  Financial Subscale | 3.10 (2.08) | 2.93 (2.02)
  News Subscale | 3.67 (1.55) | 3.66 (1.53)
  Proximity Subscale | 3.36 (1.67) | 3.41 (1.73)
  Psychological Subscale | 3.96 (1.55) | 4.13 (1.54)
  Resource Subscale: number analyzed (Participants) | 279 | 289
  Resource Subscale | 1.85 (1.17) | 1.97 (1.34)
  Symptoms Subscale | 1.57 (1.06) | 1.82 (1.24)
  Threat Subscale: number analyzed (Participants) | 279 | 289
  Threat Subscale | 4.64 (1.38) | 4.74 (1.39)

8. Secondary Outcome: Conway COVID Questionnaire Subscale Scores
Description: as for outcome 6
Time Frame: 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 280 | 289
score on a scale
  Financial Subscale | 2.91 (1.97) | 3.01 (2.07)
  News Subscale | 3.50 (1.58) | 3.67 (1.49)
  Proximity Subscale | 4.45 (1.63) | 4.56 (1.60)
  Psychological Subscale | 3.98 (1.46) | 4.18 (1.58)
  Resource Subscale | 1.81 (1.20) | 1.90 (1.27)
  Symptoms Subscale | 1.89 (1.38) | 2.13 (1.48)
  Threat Subscale | 4.81 (1.36) | 4.90 (1.33)

9. Secondary Outcome: Self-Compassion Scale Short Form Score
Description: The Self-Compassion Scale Short Form will be used to measure self-compassion. The total possible range in scores is 12-60, with higher scores indicating greater levels of self-compassion.
Time Frame: baseline, 4 weeks (post intervention), 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 342 | 315
  baseline | 35.7 (8.25) | 35.2 (8.42)
  Week 4: number analyzed (Participants) | 280 | 290
  Week 4 | 40.1 (8.75) | 36.4 (9.36)
  Week 16: number analyzed (Participants) | 280 | 289
  Week 16 | 40.3 (7.62) | 38.0 (9.28)

10. Secondary Outcome: Change From Baseline on the Perseverative Thought Questionnaire
Description: Negative ruminative thinking will be measured with the Perseverative Thought Questionnaire. The total possible range in scores is 0-60, with higher scores indicating greater levels negative ruminative thinking.
Time Frame: baseline, 4 weeks (post intervention), 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 342 | 315
  baseline | 29.89 (10.43) | 29.62 (11.29)
  Week 4: number analyzed (Participants) | 280 | 289
  Week 4 | 24.75 (10.71) | 28.19 (12.37)
  Week 16: number analyzed (Participants) | 280 | 289
  Week 16 | 23.47 (10.74) | 25.91 (12.19)

11. Secondary Outcome: Change From Baseline on the World Health Organization 5-item (WHO-5) Well-being Scale
Description: Well-being will be measured using the WHO-5. The total possible range in scores is 0-25, with higher scores indicating greater levels of well-being.
Time Frame: baseline, 4 weeks (post intervention), 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline: number analyzed (Participants) | 341 | 315
  baseline | 12.76 (4.71) | 12.47 (4.33)
  Week 4: number analyzed (Participants) | 280 | 289
  Week 4 | 15.07 (4.33) | 12.83 (4.84)
  Week 16: number analyzed (Participants) | 279 | 289
  Week 16 | 14.07 (4.64) | 12.59 (4.74)

12. Secondary Outcome: Change From Baseline on the Neutral Face Rating Task: Prosocial Construal
Description: The Neutral Face Rating task is a novel measure of prosocial construal (average likability ratings) and race bias (average liking of white faces minus the average liking of black faces). Total score for prosocial construal is from 1 to 7, with higher scores representing greater prosocial construal.
Time Frame: baseline, 4 weeks (post intervention), 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline | 4.46 (0.60) | 4.44 (0.68)
  4 weeks: number analyzed (Participants) | 281 | 291
  4 weeks | 4.42 (0.65) | 4.27 (0.59)
  16 weeks: number analyzed (Participants) | 285 | 293
  16 weeks | 4.44 (0.63) | 4.37 (0.60)

13. Secondary Outcome: Change From Baseline on the Neutral Face Rating Task: Race Bias
Description: The Neutral Face Rating task is a novel measure of prosocial construal (average likability ratings) and race bias (average liking of white faces minus the average liking of black faces). Total score for race bias range from -6 to 6, with higher scores representing greater bias favoring white faces (negative scores on the bias measure indicate bias for liking black faces more than white faces).
Time Frame: baseline, 4 weeks (post intervention), 16 weeks (3 months post-intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 344 | 318
score on a scale
  baseline | -0.57 (0.67) | -0.50 (0.68)
  4 weeks: number analyzed (Participants) | 282 | 292
  4 weeks | -0.54 (0.68) | -0.55 (0.73)
  16 weeks: number analyzed (Participants) | 285 | 293
  16 weeks | -0.51 (0.69) | -0.46 (0.67)

14. Secondary Outcome: Change From Baseline on the Growth Mindset Scale for Well-Being
Description: A measure of fixed versus incremental mindset regarding well-being. The average across items for a possible range in scores from 1-6 will be measured, with higher scores indicating greater levels of incremental views on well-being (i.e., it can be learned).
Time Frame: baseline, 4 weeks (post intervention)
Population: not all participants returned surveys for each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
Number analyzed (Participants) | 342 | 314
score on a scale
  baseline | 5.00 (0.83) | 4.94 (0.85)
  4 weeks: number analyzed (Participants) | 280 | 289
  4 weeks | 5.18 (0.81) | 4.87 (0.87)

15. Other Pre Specified Outcome: Slope Across Time on Practice Quality and Mood Items
Description: 4-tems following each app-based practice for treatment participants that ask about perceive quality of the practice, (1 poor, 9 very good), and mood (1 poor, 5 good).
Time Frame: Every other day when participant completes a practice (up to 4 weeks)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Digital Working Alliance
Description: A measure of working alliance in a digital environment that will be averaged across all items for a score range from 1 to 7, with higher scores reflecting higher levels of alliance.
Time Frame: After weeks 1, 2, and 3 during the intervention, 4 weeks (post intervention), 16 weeks (3 months post-intervention) - Intervention group only
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Description: Anxiety and depression scores were characterized separately at T1 (baseline), T5 (4 weeks), and T6 (16 weeks) based on normative none-to-slight, mild, moderate, and severe symptoms from PROMIS anxiety and PROMIS depression scores (i.e., T-score <55, 55≥ <60, 60≥ <70, and ≥70; Pilkonis et al., 2011).
Arm/Group | Healthy Minds Program Foundations Training | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/344 | 0/318
Serious Adverse Events (participants affected / at risk) | 0/344 | 0/318
Other Adverse Events (participants affected / at risk) | 344/344 | 318/318
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Minds Program Foundations Training (N=344) | Wait-list Control (N=318)
None to Slight Depression at Baseline (Nervous system disorders) | 175 | 160
Mild Depression at Baseline (Nervous system disorders) | 80 | 65
Moderate Depression at Baseline (Nervous system disorders) | 87 | 87
Severe Depression at Baseline (Nervous system disorders) | 1 | 3
None to Slight Depression at 4 weeks (Nervous system disorders) | 218 | 172
Mild Depression at 4 weeks (Nervous system disorders) | 36 | 51
Moderate Depression at 4 weeks (Nervous system disorders) | 25 | 61
Severe Depression at 4 weeks (Nervous system disorders) | 1 | 5
None to Slight Depression at 16 weeks (Nervous system disorders) | 205 | 171
Mild Depression at 16 weeks (Nervous system disorders) | 46 | 57
Moderate Depression at 16 weeks (Nervous system disorders) | 30 | 61
Severe Depression at 16 weeks (Nervous system disorders) | 1 | 1
None to Slight Anxiety at Baseline (Nervous system disorders) | 77 | 69
Mild Anxiety at Baseline (Nervous system disorders) | 98 | 99
Moderate Anxiety at Baseline (Nervous system disorders) | 154 | 130
Severe Anxiety at Baseline (Nervous system disorders) | 14 | 17
None to Slight Anxiety at 4 weeks (Nervous system disorders) | 133 | 91
Mild Anxiety at 4 weeks (Nervous system disorders) | 75 | 80
Moderate Anxiety at 4 weeks (Nervous system disorders) | 69 | 105
Severe Anxiety at 4 weeks (Nervous system disorders) | 3 | 13
None to Slight Anxiety at 16 weeks (Nervous system disorders) | 113 | 100
Mild Anxiety at 16 weeks (Nervous system disorders) | 89 | 80
Moderate Anxiety at 16 weeks (Nervous system disorders) | 79 | 96
Severe Anxiety at 16 weeks (Nervous system disorders) | 1 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT04426318/Prot_SAP_000.pdf